CLINICAL TRIAL: NCT02520973
Title: Screening for TB in Pregnancy A Supplement to: The Effect of Tuberculosis and Its Treatment on HIV-Infected Pregnant Women and Their Infants
Brief Title: Screening for TB in Pregnancy. on HIV-Infected Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 00039194
Record Dates: First submitted 2015-03-09; First posted 2015-08-13 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Universal screening (Experimental): All HIV + pregnant women will be asked to give a sputum sample for TB prior to TB symptom screen
  Interventions: Other: Sputum sample
- Symptom- directed screening (Active Comparator): Only symptomatic HIV+ pregnant women will be asked to give a sputum sample for TB
  Interventions: Other: Sputum sample

INTERVENTIONS:
Other: Sputum sample

SUMMARY:
Pregnant women who develop active Tuberculosis (TB) are at increased risk of poor maternal and infant outcomes. Our data from South Africa show that up to 3% of HIV-infected pregnant women have active TB , many with advanced disease, contributing to the 40% of maternal mortality associated with TB or HIV in South Africa . Screening for TB in pregnant women in this setting is therefore essential to reduce maternal mortality. Symptom-directed screening for TB has been recommended by the World Health Organization and by the South African National Department of Health; however, no implementation framework is in place to operationalize the guidelines. Symptom-based testing is an efficient process that limits use of diagnostic tests, but may miss many cases. In Soweto, we found that 0.7% (700/100,000) of HIV-infected women had active TB when a symptom-based strategy was employed once, but in Klerksdorp we found that 3.3% (3,300/100,000) had active TB when universal testing, regardless of symptoms, was performed; most TB cases were newly diagnosed among women who reported no symptoms .

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositive by two rapid tests, or documented history of a positive Enzyme Immunoassay EIAs, or HIV RNA >1000 copies/mL
2. Pregnancy confirmed by urine pregnancy test or clinical exam
3. Estimated gestational age of 13 weeks or older
4. Age 18 years or greater
5. Willing to provide verbal consent

Exclusion Criteria:

1. Currently diagnosed with TB
2. Completed TB treatment within the last 6 months
3. Inability to communicate in one of the study languages.
4. Lack of comprehension of the study based on inability to meet basic understanding questions during the screening process.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women diagnosed with TB | One year
  1. Proportion of women who are diagnosed with TB in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chaisson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Perinatal HIV Research Unit, Klerksdorp, Northwest, South Africa